CLINICAL TRIAL: NCT03991221
Title: Validation of Schematic Representations for Dental Malocclusion and Craniofacial Deformities Screening in Temporary and Mixed Dentition Requiring Early Orthodontic Treatment
Brief Title: Validation of Dental Malocclusion Schematic Representations for Early Orthodontic Treatment
Acronym: CHARTE-ODF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: APHP180562; 2019-A01074-53 (Other: IDRCB)
Record Dates: First submitted 2019-05-24; First posted 2019-06-19 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Dental Malocclusion
Keywords: Prevention; Early treatment; Skeletal discrepancy; Malocclusion
MeSH Terms: conditions — Malocclusion | interventions — Diagnosis, Oral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental exam by orthodontic non-specialists (Other): Detection of the presence of at least one malocclusion by orthodontic non-specialists with the graphic chart
  Interventions: Other: Dental Exam
- Dental exam by orthodontic experts (Other): Detection of the presence of at least one malocclusion by orthodontic experts
  Interventions: Other: Dental Exam; Other: Orthodontics consult; Other: Call back at 6 month

INTERVENTIONS:
Other: Dental Exam — Visual examination of the child oral cavity bi non-orthodontist experts and orthodontist expert
Other: Orthodontics consult — Consultation with an orthodontics specialist if a malocclusion requiring early intervention is detected
  Arms: Dental exam by orthodontic experts
Other: Call back at 6 month — Telephone call back at six months of inclusion in the study if a malocclusion requiring early intervention is detected
  Arms: Dental exam by orthodontic experts

SUMMARY:
Dental occlusion is the reciprocal confrontation of the two dental arches. The child has two set of temporary and permanent teeth and passes through different stages of dentition during which dental, skeletal or functional abnormalities may appear.

Dental malocclusion is defined as an incorrect position of the teeth in the bone base, as well as the incoordination of the teeth of the opposite arches or the displacement of the maxillary and mandibular skeletal bases.

When a malocclusion is detected during clinical examination, patients are referred to an orthodontic specialist. The interception in orthodontics is carried out during a growing period; it consists of correcting or reducing malocclusions in evolution and eliminating the functional causes to prevent aggravation of skeletal and dental abnormalities.

An epidemiological study conducted in France on 789 children showed that 37.4% had at least one type of dental malocclusion. In 2010, a study of 5988 French children showed that 14% of them had received orthodontic treatment. These studies reveal a discrepancy between treatment needs and treatments conducted. In addition, certain dental malocclusions and skeletal disorders, such as lateral and anterior crossbite, require early orthodontic treatment in order to avoid aggravation of the occlusion disorder and induction of craniofacial growth disorders. Unfortunately these discrepancies are not always detected by the caregivers (pediatrician, general dentist, pediatric dentist).

A schematic representation of malocclusions in temporary and mixed dentition requiring orthodontic interception has been developed by the investigator's team to provide a simple visual means of identifying these dental and skeletal disorders in order to improve early screening by practitioners involved in the mandatory medical follow-up of children.

DETAILED DESCRIPTION:
Dental malocclusion is defined as an incorrect position of the teeth in the bone base, as well as the incoordination of the teeth of the opposite arches or the displacement of the maxillary and mandibular skeletal bases.

When a malocclusion is detected during clinical examination, patients are referred to an orthodontic specialist. The interception in orthodontics is carried out during a growing period; it consists of correcting or reducing malocclusions in evolution and eliminating the functional causes to prevent aggravation of skeletal and dental abnormalities. Early intervention is critical for specific dental malocclusions and skeletal disorders, such as lateral and anterior crossbite in order to avoid aggravation of the occlusion disorder and induction of craniofacial growth disorders. Unfortunately these discrepancies are not always detected by the caregivers (pediatrician, general dentist, pediatric dentist).

ELIGIBILITY:
Inclusion Criteria:

* child between 5 and 10 years old
* seen in consultation with pediatrician, pediatric dentist, or general dentist,

Exclusion Criteria:

* child not letting himself be examined,
* children who have already received orthodontic treatment and / or are currently undergoing orthodontic treatment
* Absence of free and informed consent
* Non affiliation to a social security regime or CMU

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 659 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Detection the presence of at least one malocclusion in children, requiring an early orthodontic treatment, compared to orthodontic experts (gold-standard) | 2 months
  Study of the performance of orthodontic non-specialists with the graphic chart to detect the presence of at least one malocclusion in children, requiring an early orthodontic treatment, compared to orthodontic experts (gold-standard)

SECONDARY OUTCOMES:
Detection of each type of malocclusion requiring early orthodontic treatment by non-orthodontist practitioners versus orthodontic experts | 2 months
Prevalence of malocclusions identified by orthodontic experts | 2 months
Number of orthodontic consultations within 6 months among children screened for a malocclusion reacquiring early orthodontic treatment | 6 months
Number of orthodontic treatments started within 6 months among children screened for a malocclusion reacquiring early orthodontic treatment | 6 months

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Hôpital de jour pédiatrique - Hôpital Louis Mourier, Colombes
  - Odontologie Pédiatrique - Hôpital Louis Mourier, Colombes
  - Servide d'odontologie - Hôpital Louis Mourier, Colombes
  - Endocrinologie et diabète de l'enfant - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Neurologie Pédiatrique - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Cabinet d'odontologie pédiatrique, Montrouge
  - Cabinet privé pédiatrique, Paris
  - Cabinet privé pédodontie, Paris
  - Odontologie Pédiatrique - Hôpital Bretonneau, Paris
  - Service d'odontologie - Hôpital Bretonneau, Paris
  - Cabinet privé d'odontologie, Paris